CLINICAL TRIAL: NCT07342972
Title: Effect of a Goat-milk Based Infant Formula on Gastrointestinal Symptoms and Tolerability in Healthy Term Infants: a Double-blind Randomized Controlled Trial
Brief Title: Gastrointestinal Symptoms and Tolerance in Infants Fed Goat or Cow's Milk-based Infant Formula
Acronym: MESK-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ausnutria Hyproca B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P24-150
Record Dates: First submitted 2025-12-23; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Tolerance; Gastrointestinal Symptoms; Infections; Quality of Life; Anthropometrics
Keywords: Formula; Infant; Goat milk-based infant formula; RCT; Gastrointestinal symptoms; Gastrointestinal tolerance
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double-blind clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Goat milk-based infant formula
  Interventions: Other: Goat milk-based infant formula
- Control group (Active Comparator): Cow's milk-based infant formula
  Interventions: Other: Cow's milk-based infant formula

INTERVENTIONS:
Other: Goat milk-based infant formula — Study product is administered on demand until the age of 6 months.
  Arms: Intervention group
Other: Cow's milk-based infant formula — Study product is administered on demand until the age of 6 months.
  Arms: Control group

SUMMARY:
This randomized controlled double-blind study will compare the effect of a commercially available goat milk formula to a cow's milk formula on gastrointestinal symptoms and tolerance, and infections in infants.

ELIGIBILITY:
Inclusion Criteria:

* Age between 14 days and 90 days.
* Healthy singleton term infants born between 37 weeks and 42 weeks of gestation.
* Infants who have received CMF for at least 7 consecutive days.
* Exclusive formula feeding.
* Cow's Milk-related Symptoms Score (CoMiSS®) value at baseline of ≥6 and <10.
* Parents' or caregivers, aged ≥18 years, willing to give informed consent and adhere to study protocol

Exclusion Criteria:

* Exclusively or partially feeding with human milk
* Introduced to solid food, supplementary feeding, use of pre- and/or probiotics as a supplement
* Congenital or recurrent chronic conditions and/or malabsorption that could interfere with study parameters.
* Diagnosed cow's milk allergy (CMA) or suspected to have CMA, soy allergy, fish allergy, egg allergy and/or lactose intolerance.
* Receiving medication (on own initiative or prescription) with regard to FGID (i.e. reflux medication)
* Sibling already participating in this study
* Participation in another clinical trial

Ages: 14 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal symptoms as determined by CoMiSS | Difference between groups at Day 14 of the intervention
  The CoMiSS® is a simple, fast, and easy-to-use awareness tool for cow's milk-related symptoms and may be used in clinical trials to evaluate and quantify the severity of symptoms during a feeding trial. The CoMiSS scores symptoms in five different domains: Crying, Regurgitation, Stools, Skin and Respiratory. The CoMiSS score ranges from 0 to 33 with score 0 as best score (no symptoms) and 33 as worst score (severe symptoms).
Gastrointestinal tolerance as determined by IGSQ | Difference between groups at the end of the intervention at 24 weeks
  The IGSQ is a 13-item self-report instrument that has been used in clinical trials to assess infants' GI-related signs and symptoms observed by their parents over the previous week in 5 domains: stooling, regurgitation/vomiting, flatulence, crying, and fussiness. The IGSQ has a possible range of 13 to 65, where higher values indicate greater GI distress and values ≤ 23 indicate no digestive distress.

SECONDARY OUTCOMES:
Gastrointestinal symptoms throughout the study as determined by CoMiSS | From enrollment to the end of the intervention at 24 weeks
  The CoMiSS® is a simple, fast, and easy-to-use awareness tool for cow's milk-related symptoms and may be used in clinical trials to evaluate and quantify the severity of symptoms during a feeding trial. The CoMiSS scores symptoms in five different domains: Crying, Regurgitation, Stools, Skin and Respiratory. The CoMiSS score ranges from 0 to 33 with score 0 as best score (no symptoms) and 33 as worst score (severe symptoms).
Gastrointestinal tolerance throughout the study as determined by IGSQ | From enrollment to the end of the intervention at 24 weeks
  The IGSQ is a 13-item self-report instrument that has been used in clinical trials to assess infants' GI-related signs and symptoms observed by their parents over the previous week in 5 domains: stooling, regurgitation/vomiting, flatulence, crying, and fussiness. The IGSQ has a possible range of 13 to 65, where higher values indicate greater GI distress and values ≤ 23 indicate no digestive distress.
Occurrence, duration and severity of gastrointestinal infections as determined by Vesikari | From enrollment to the end of the intervention at 24 weeks
  The Vesikari Clinical Severity Scoring System includes a e-diary card completed by parents, to identify rotavirus gastroenteritis episodes. The Vesikari Clinical Severity Scoring System Parameters score ranges from 0 to 20 with score <7 as mild symptoms and score 10 to 20 as severe symptoms.
Occurrence, duration and severity of respiratory infections as determined by CARIFS | From enrollment to the end of the intervention at 24 weeks
  Canadian Acute Respiratory Illness and Flu Scale is a validated parental questionnaire, to measure the disease severity of children with acute respiratory illness (ARI) including influenza. CARIFS consists of 18 items covering three domains; symptoms (e.g., cough); function (e.g., play), and parental impact (e.g., clinginess). Each item is scored 0 to 3, with higher scores indicating greater severity of illness. The full scale ranges from 0 to 58. For children older than 5 years the full scale is used; for children younger than 5 years, 3 items (headache, sore throat, and muscle aches) are not used for assessment.
Occurrence, duration and severity of ear infections as determined by AOM-SOS V5 | From enrollment to the end of the intervention at 24 weeks
  The Acute Otitis Media Symptom Severity scale (AOM-SOS) Version 5.0 is psychometric scale used to measure the severity of symptoms in children with acute otitis media and has been validated for parent-reported use. A 6-point Likert scale ranging from 'No' to 'An extreme amount' is used to rate the presence of 5 symptoms related to acute otitis media over the preceding 24 hours. The AOM-SOS Version 5.0 total score is obtained by summing the scores on these 5 equally-weighted questions.
Quality of life as determined by PedsQL | From enrollment to the end of the intervention at 24 weeks
  The Pediatric Quality of Life Inventory (PedsQL™) Infant Scales™ is a specific module of the PedsQL™. The objective of this validated questionnaire is to measure generic health-related quality of life in infants. Applicable for infants with acute and chronic health conditions and healthy infants. The questionnaire is composed of 36 items comprising 5 dimensions: physical functioning, physical symptoms, emotional functioning, social functioning and cognitive functioning. Higher scores means better HRQOL and fewer problems or symptoms. A 5-point Likert scale from is applied: 0 (Never) to 4 (Almost always). Scores are transformed on a scale from 0 to 100.
Quality of life as determined by WHOQoL-BREF | From enrollment to the end of the intervention at 24 weeks
  The World Health Organization Quality of Life Questionnaire BREF (WHOQoL-BREF) is the shortened version of the WHOQoL-100. The WHOQoL-BREF measures quality of life within the context of an individual's culture, value systems, personal goals, standards of concerns. The measuring instrument consists of 26 items. The raw scoreis transformed to a 0-100 scale, where higher scores indicate higher perceived quality of life.
Weight | From enrollment to the end of the intervention at 24 weeks
  Weight will be measured in kilograms.
Height | From enrollment to the end of the intervention at 24 weeks
  Height will be measured in centimeters.
Head circumference | From enrollment to the end of the intervention at 24 weeks
  Head circumference will be measured in centimeters.
WHO z-scores | From enrollment to the end of the intervention at 24 weeks
  Subject's weight, length and head circumference will be used to calculate the WHO z-scores for weight-for-age, length-for-age, head circumference-for-age, weight-for-length.
Fecal parameters | Baseline, Day 14, Day 28, Week 12 and Week 24
  The major fecal bacterial groups are defined using 16S RNA sequencing. Further fecal parameters (e.g. pH, SCFA, sIgA, A1AT) are determined with standard laboratory techniques.
Sleep and Crying episodes | Baseline, Day 14, Day 28, Week 12 and Week 24
  Sleep and crying episodes and duration are recorded for 24 hours prior to the visits in diaries.
Stool frequency & consistenty | Baseline, Day 14, Day 28, Week 12 and Week 24
  Stool frequency and consistency are recorded for 24 hours prior to visits in diaries.

CONTACTS AND LOCATIONS:
Locations (1):
- King Faissal Specialist Hospital & Research Centre, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No